CLINICAL TRIAL: NCT00005394
Title: Diagnosis/Pathophysiology of Glucocorticoid Remediable Aldosteronism Hypertension
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4300; R01HL053693 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Hypertension; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Heart Diseases

SUMMARY:
To identify and study a large cohort of glucocorticoid remediable aldosteronism (GRA) patients.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

The spectrum of the severity and the natural history of the disorder was characterized. Modifying environmental and genetic factors important in regulation of blood pressure were determined. Also, renal physiology was studied in GRA patients to determine how these patients escaped hypokalemia in spite of mineralocorticoid excess. There were four specific aims including: 1) to determine the natural history and prevalence of GRA in various hypertensive populations, 2) to characterize the magnitude of effect imparted on blood pressure by inheritance of GRA and the sources of variation in phenotype expression of the hypertension, 3) to investigate the renal and hormonal mechanisms regulating potassium conservation and loss in GRA, and 4) to characterize the disequilibrium of GRA with Irish and Scottish descent and specific alleles of the aldosterone synthase gene.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-08; Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lifton — Yale University

REFERENCES:
- [Background] Litchfield WR, Coolidge C, Silva P, Lifton RP, Fallo F, Williams GH, Dluhy RG. Impaired potassium-stimulated aldosterone production: a possible explanation for normokalemic glucocorticoid-remediable aldosteronism. J Clin Endocrinol Metab. 1997 May;82(5):1507-10. doi: 10.1210/jcem.82.5.3964. PMID 9141541
- [Background] Litchfield WR, Anderson BF, Weiss RJ, Lifton RP, Dluhy RG. Intracranial aneurysm and hemorrhagic stroke in glucocorticoid-remediable aldosteronism. Hypertension. 1998 Jan;31(1 Pt 2):445-50. doi: 10.1161/01.hyp.31.1.445. PMID 9453343
- [Background] Litchfield WR, New MI, Coolidge C, Lifton RP, Dluhy RG. Evaluation of the dexamethasone suppression test for the diagnosis of glucocorticoid-remediable aldosteronism. J Clin Endocrinol Metab. 1997 Nov;82(11):3570-3. doi: 10.1210/jcem.82.11.4381. PMID 9360508